CLINICAL TRIAL: NCT02980393
Title: The Impact of a Structured Lifestyle Intervention on Body Composition and Exercise Capacity in Overweight Children With Operated Heart Defects
Brief Title: Smart Heart Trial: Structured Lifestyle Intervention for Overweight and Obese Youth With Operated Heart Defects
Acronym: SHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kambiz Norozi (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Kambiz Norozi, Paediatric Cardiologist, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 102392; 18843 (Other: UWesternOntario)
Record Dates: First submitted 2016-11-24; First posted 2016-12-02 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Congenital Heart Disease; Pediatric Obesity
Keywords: congenital heart disease; smart mobile technology; children; adolescents; lifestyle counselling; nutrition; physical activity
MeSH Terms: conditions — Heart Defects, Congenital; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle intervention (Experimental): Participants are guided by a fitness specialist who will help the participants to incorporate physical activity into their daily life. Based on the cardiologist assessment, an individual home-based exercise program will be developed. Participants are also guided and advised on nutrition with emphasis on low fat content and increased fiber. The nutrition counseling will focus on sustainable changes and will help participants to make healthy food choices.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — The structured lifestyle intervention involves alternating weekly phone calls with two health coaches: a registered dietitian and a fitness specialist. A total of 50 phone calls (25 nutrition-related and 25 physical activity-related) are delivered over the one-year study. After six months in the program, participants are introduced to supporting program-specific software that they can access online, as an additional way to interact with the program, set goals, and record their progress. Client and family-centred nutrition and physical activity counselling includes an initial and regular behavioural assessment, and subsequent conversations (i.e., phone calls) using motivational interviewing techniques intended to increase knowledge or skills, and improve behaviours.

SUMMARY:
This study is to assess whether a lifestyle intervention with diet, exercise and counselling in young patients will have a positive influence on their weight and overall well-being. This study will enrol patients between the ages of 7 to 17 years of age, who have congenital heart disease, and have been identified being overweight or obese. A total of 40 individuals will participate in this study. The study duration will last for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* overweight or obese (BMI> 85%) patients
* between 7-17 years of age
* operated or non-operated congenital heart disease
* reside in Southwestern Ontario

Exclusion Criteria:

* inability to comply with research testing or intervention components due to mental and/or physical disabilities, medications or comorbidities affecting weight or metabolic condition
* involvement in any concurrent lifestyle intervention program

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Baseline Body Mass Index (BMI) at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  BMI is derived from body mass divided by the square of the body height
Change in Baseline Fat Mass at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Dual energy x-ray absorptiometry (DEXA) will measure fat mass.
Change in Baseline Lean Mass at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Dual energy x-ray absorptiometry (DEXA) will measure lean mass.
Change in Baseline Percent Fat at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Dual energy x-ray absorptiometry (DEXA) will measure percent fat.
Change in Baseline Percent Android Fat at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Dual energy x-ray absorptiometry (DEXA) will measure percent android fat.
Change in Baseline Visceral Adipose Tissue at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Dual energy x-ray absorptiometry (DEXA) will measure visceral adipose tissue.
Change in Baseline Bone Mineral Content at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Dual energy x-ray absorptiometry (DEXA) will measure bone mineral content.
Change in Baseline Maximum Oxygen Consumption at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Maximal exercise graded treadmill test will determine maximal oxygen consumption.

SECONDARY OUTCOMES:
Change in Baseline Average Caloric Intake at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Average caloric intake is estimated from three-day food records.
Change in Baseline Self-Report Physical Activity Levels at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Physical activity levels will also be measured by the Physical Activity Questionnaire for Older Children
Change in Baseline Physical Activity Levels at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Physical activity levels will be measured from accelerometers
Change in Baseline Quality of Life at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Pediatric Quality of Life Inventory Generic Core Scales
Change in Baseline Muscle function at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Leonardo Mechanograph® Ground Reaction Force Plate will assess jumping height.
Change in Baseline Electrocardiographic measurement at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Electrocardiogram
Change in Baseline Transthoracic echocardiographic measurement at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Echo-cardiogram will be employed.
Change in Baseline Endothelial vasodilator function at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Peripheral arterial tonometry will assess endothelial vasodilator function.
Change in Baseline Lipid Profile at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Blood is drawn from patients who have been asked to fast for at least 10 hours.
Change in Baseline Electrolytes at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Blood is drawn from patients who have been asked to fast for at least 10 hours.
Change in Baseline Creatinine at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Blood is drawn from patients who have been asked to fast for at least 10 hours.
Change in Baseline Urea at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Blood is drawn from patients who have been asked to fast for at least 10 hours.
Change in Baseline Fasting Glucose at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Blood is drawn from patients who have been asked to fast for at least 10 hours.
Change in Baseline Serum Insulin at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Blood is drawn from patients who have been asked to fast for at least 10 hours.
Change in Baseline Adiponectin at 1 year | This outcome was measured at Baseline, 6 months, 1 year within the 1 year time frame
  Blood is drawn from patients who have been asked to fast for at least 10 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz Norozi, MD, PhD, Principal Investigator — London Health Science Centre

REFERENCES:
- [Derived] Rombeek M, De Jesus S, Altamirano-Diaz L, Welisch E, Prapavessis H, Seabrook JA, Norozi K. The use of smartphones to influence lifestyle changes in overweight and obese youth with congenital heart disease: a single-arm study: Pilot and feasibility study protocol: Smart Heart Trial. Pilot Feasibility Stud. 2017 Nov 15;3:59. doi: 10.1186/s40814-017-0207-y. eCollection 2017. PMID 29167745